CLINICAL TRIAL: NCT06048042
Title: Clinical and Radiographic Evaluation of Autogenous Demineralized Dentin Graft Versus Autogenous Bone Graft in Management of Periodontal Intrabony Defects Using Modified Minimally Invasive Surgical Technique: A Non-Randomized Clinical Trial
Brief Title: Evaluation of Autogenous Demineralized Dentin Graft Vs Autogenous Bone Graft in Management of Intrabony Defects
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ghada Mohamed Ali Hussein Abouhussein, Master Degree student, Periodontology department, Faculty of Dentistry, Cairo University, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ghadashatra123
Record Dates: First submitted 2023-09-09; First posted 2023-09-21 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Intrabony Periodontal Defect
Keywords: Intrabony Periodontal Defect; Demineralized dentin graft; Autogenous bone graft; modified minimally invasive surgical technique; M-MIST

STUDY DESIGN:
Intervention Model Description: A non-randomized Clinical Trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autogenous Demineralized Dentin Graft (Experimental): An Autogenous Demineralized Dentin Graft will be prepared from the participant's freshly extracted teeth and placed in the intrabony defect following the modified minimally invasive surgical technique.
  Interventions: Biological: Autogenous Demineralized Dentin Graft
- Autogenous bone Graft (Active Comparator): An Autogenous Bone Graft will be harvested from the retromolar area and placed in the intrabony defect following the modified minimally invasive surgical technique.
  Interventions: Biological: Autogenous Bone Graft

INTERVENTIONS:
Biological: Autogenous Demineralized Dentin Graft — The participant's own freshly extracted tooth will be cleaned from periodontal ligaments, cementum, soft tissue attachment, caries, or restorations (if present) and have their crown decapitated, using a high- speed fine finishing stone and saline irrigation. The pulp chamber and root pulp will be cleaned by split opening the root and cleaning it out using a high-speed diamond bur. Subsequently, teeth will be ground, and demineralized using a hand bone mill. Then the particles will be prepared by demineralization of tooth particles in 0.6N hydrochloric acid5 for 30 min then washed twice in saline and dried with sterile gauze. Then it will be used as a graft for the intra-bony defect after modified minimally invasive surgical technique.
  Arms: Autogenous Demineralized Dentin Graft
Biological: Autogenous Bone Graft — Modified minimally invasive surgical technique (M-MIST) will be performed in the intra-bony defects, with autogenous bone graft placement. The graft will be harvested from the retromolar area using automatic chip maker (ACM) bur and a hand bone mill will be used to grind the chips into particles, then it will be placed in the defect.
  Arms: Autogenous bone Graft

SUMMARY:
The main goal is to evaluate and compare the clinical and radiographic efficacy of autogenous demineralized dentin as bone graft substitute versus autogenous bone graft when performed with modified minimally invasive surgical technique (M-MIST) in the treatment of periodontal intrabony defects.

The main question is: In periodontitis patients with intrabony defects, will using autogenous demineralized dentin as bone graft substitute result in clinical attachment gain and linear bone fill similar to autogenous bone graft following modified minimally invasive surgical technique? After enrolment, each participant with intra-bony defects will receive the initial phase of the therapy, which will include oral hygiene instructions, supragingival and subgingival debridement using ultrasonic and hand instrumentations and relieving of occlusal trauma if any.

After 4-6 weeks, an individually customized positioning stent will be fabricated for each participant and a pre-operative periapical x-ray using parallel-angle technique will be employed using X-ray film holding system to ensure accuracy and reproducibility of the measurements.

Criteria used to indicate that surgery is required include the persistence of interproximal defect with PD (Probing depth) ≥ 5 mm, CAL (Clinical attachment loss) ≥ 4 mm.

Surgical procedures will include flap elevation for approaching the defect-associated sites using the modified minimally invasive surgical technique (M-MIST).

Intervention group: The defect will be filled with autogenous demineralized dentin graft prepared from the participant's freshly extracted own teeth.

Control group: The defect will be filled with autogenous bone graft harvested from the retromolar area.

For both groups, flaps will be approximated and sutured at the original position. All the subjects will be evaluated at 1, 3, and 6 months for clinical and radiographic parameters. Outcomes:The results of Clinical attachment level (CAL) gain, Linear bone fill, Gingival index (GI), Plaque index (PI), Probing pocket depth (PPD), Gingival recession (GR), Bleeding on probing (BoP), Postoperative pain and Patient satisfaction will be measured at baseline, 1 month, 3 months and after 6 months.

DETAILED DESCRIPTION:
Research objective: The aim of conducting this research is the development of a newer, less invasive and cost-effective therapeutic approaches that help in management of periodontal intrabony defects. Due to the shortcomings of other bone substitute materials, another bone substitute material that would be completely autogenous and cost-effective is required. Grafting autogenous demineralized dentin has been used extensively for socket preservation and showed promising results in addition to being cost-effective.

Research Procedure in brief:

This study will be carried out on patients enrolled from the Outpatient Clinic of Oral Medicine and Periodontology department, Faculty of Dentistry, Cairo University.

Eligibility criteria:

I. Inclusion criteria:

Patient-related criteria:

* Motivated patient 18 years of age or order.
* Patient consulting in the outpatient clinic.
* Patient ready to perform oral hygiene instructions.
* Provide informed consent.
* Accepts the 6 months follow-up period.

Teeth related criteria:

* Tooth with two or three-walled intra-bony defect, probing depth ≥ 5mm with intra osseous defect ≥ 3mm.
* Mature permanent tooth.
* Unrestorable tooth or fractured tooth beyond restoration, impacted third molar or supernumerary tooth to be extracted and used as whole tooth graft inside the intrabony defect.

II. Exclusion criteria:

Patient-related criteria:

* Medically compromised patients.
* Pregnant women.
* Uncooperative patients.
* Smokers.
* Systemic diseases that may compromise healing or bone metabolism (e.g diabetes, hyperthyroidism).
* Failure to maintain good oral hygiene.

Teeth related criteria:

* Teeth with supra-bony defects.
* Teeth with grade III mobility.
* Teeth having interproximal craters, grade III furcation involvement, and grade III mobility.
* Presence of caries or overhanging restorations.
* Presence of peri-apical injuries.

General operative procedure:

* The selected participants will be informed about the nature of the research and its procedures, then written informed consent will be obtained.
* The surgical procedure will be explained to all patients prior to surgery.
* Patients diagnosed with periodontitis who meet the inclusion criteria will be screened for periodontal examination. Based on this examination, target sites will be identified.
* Each patient will receive the initial phase of the therapy, which will include oral hygiene instructions, supragingival and subgingival debridement using ultrasonic and hand instrumentations and relieving of occlusal trauma if any.

Pre-surgical patient preparation (Re-evaluation phase):

* 4-6 weeks after the initial therapy, periodontal re-evaluation will be done to confirm the sites that will require surgical therapy.
* Criteria used to indicate that surgery is required include the persistence of interproximal defect with PD ≥ 5 mm, CAL ≥ 4 mm.
* An individually customized positioning stent will be fabricated for each patient and a pre-operative periapical x-ray using parallel-angle technique will be employed using X-ray film holding system to ensure accuracy and reproducibility of the measurements.
* A periapical radiograph using paralleling technique using KCP film holder will be performed for each patient to evaluate alveolar bone loss using DIGORA system.

Surgical procedures

* Pre-procedural mouth rinse using 0.2% chlorhexidine gluconate3 rinses for intraoral antisepsis.
* Surgical sites will be anaesthetized using local anesthesia4.
* The defect-associated inter-dental papilla will be surgically approached either with a diagonal incision following the pattern of the simplified papilla preservation flap when the width of the inter-dental space is 2 mm or narrower or with a horizontal incision according to the modified papilla preservation technique at inter-dental sites wider than 2 mm.
* Flap elevation will be limited to the buccal flap.
* No inter-dental and/or lingual intra-sulcular incisions will be performed.
* After removal of the granulation tissue by careful dissection and root debridement, the root surface will be chemically conditioned with a 2 min. application of an EDTA gel.

The participants will be divided into two groups:

Intervention group:

• The participant's own freshly extracted tooth will be cleaned from periodontal ligaments, cementum, soft tissue attachment, caries, or restorations (if present) and have their crown decapitated, using a high- speed fine finishing stone and saline irrigation. The pulp chamber and root pulp will be cleaned by split opening the root and cleaning it out using a high-speed diamond bur. Subsequently, teeth will be ground, and demineralized using a hand bone mill. Then the particles will be prepared by demineralization of tooth particles in 0.6N hydrochloric acid5 for 30 min then washed twice in saline and dried with sterile gauze. Then it will be used as a graft for the intra-bony defect after modified minimally invasive surgical technique.

Control group:

* Modified minimally invasive surgical technique (M-MIST) will be performed in the intra-bony defects, with autogenous bone graft placement. The graft will be harvested from the retromolar area using automatic chip maker (ACM) bur and a hand bone mill will be used to grind the chips into particles, then it will be placed in the defect.
* For both groups, flaps will be approximated and sutured at the original position with a 5-0 monofilament polypropylene suture material using simple direct loop interrupted technique.

Post-operative care and follow-up

* Participants will be instructed to abstain from trauma on the operative site, not to interfere with the suture and to avoid hot food or vigorous rinsing.
* Tooth brushing will be encouraged for other parts of the dentition and gentle tooth brushing for the operative site will be advised to be resumed after two weeks.
* Participants will be prescribed Ibuprofen 600 mg.
* Chlorhexidine 0.12% mouthwash will be prescribed for gentle rinsing twice daily for two weeks.
* Sutures will be removed two weeks after the surgery.
* All the subjects will be evaluated at 1, 3, and 6 months for clinical and radiographic parameters. Outcomes:The results of Clinical attachment level (CAL) gain, Linear bone fill, Gingival index (GI), Plaque index (PI), Probing pocket depth (PPD), Gingival recession (GR), Bleeding on probing (BoP), Postoperative pain and Patient satisfaction will be measured at baseline, 1 month, 3 months and after 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient-related criteria:

  * Motivated patient 18 years of age or order.
  * Patient consulting in the outpatient clinic.
  * Patient ready to perform oral hygiene instructions.
  * Provide informed consent.
  * Accepts the 6 months follow-up period.
* Teeth related criteria:

  * Tooth with two or three-walled intra-bony defect, probing depth ≥ 5mm with intra osseous defect ≥ 3mm.
  * Mature permanent tooth.
  * Unrestorable tooth or fractured tooth beyond restoration, impacted third molar or supernumerary tooth to be extracted and used as whole tooth graft inside the intrabony defect.

Exclusion Criteria:

* Patient-related criteria:

  * Medically compromised patients.
  * Pregnant women.
  * Uncooperative patients.
  * Smokers.
  * Systemic diseases that may compromise healing or bone metabolism (e.g diabetes, hyperthyroidism).
  * Failure to maintain good oral hygiene.
* Teeth related criteria:

  * Teeth with supra-bony defects.
  * Teeth with grade III mobility.
  * Teeth having interproximal craters, grade III furcation involvement, and grade III mobility.
  * Presence of caries or overhanging restorations.
  * Presence of peri-apical injuries.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-07-17 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Clinical attachment level (CAL) gain change from baseline to 6 months. | CAL gain will be taken at baseline, 1 month, 3 months and 6 months after the intervention during the follow-up period and will be done by a single calibrated examiner.
  The CAL will be clinically measured using UNC 15 periodontal probe from the cemento-enamel junction (CEJ) to the depth of defect. An individually customized positioning stent will be fabricated for each patient to ensure accuracy and reproducibility of the measurements.

SECONDARY OUTCOMES:
Linear bone fill change from baseline to 6 months | Linear bone fill will be measured at baseline, 3 months and 6 months after the intervention during the follow-up period and will be done by a single calibrated examiner
  Linear bone fill will be radiographically measured from the CEJ to the deepest part of the intrabony defect using the linear measurement tool of the Digora software. Individually customized positioning stent will be fabricated for each patient and parallel-angle technique will be employed using X-ray film holding system. This will ensure accuracy and reproducibility of the measurements. Radiographic linear defect depth (RLDD) will be measured as the depth of the intrabony defect from the alveolar crest to the defect base at baseline and 6 months postoperatively. The defect angle will be measured at baseline, as the angle formed between intersections of lines from the alveolar crest to the defect base and tooth long axis line. Calculation of bone fill in mm will be done by a subtraction of follow-up from baseline RLDD values, and percentages of bone fill will be expressed as the proportion of change to baseline RLDD.
Gingival index (GI) change from baseline to 6 months | GI will be measured baseline, 1 month, 3 months and 6 months after the intervention during the follow-up period and will be done by a single calibrated examiner
  The GI will be evaluated by using Silness-Loe GI (0 = Normal gingiva, 1 = Mild inflammation, 2 = Moderate inflammation, 3 = Severe inflammation).
Plaque index (PI) change from baseline to 6 months | PI will be measured baseline, 1 month, 3 months and 6 months after the intervention during the follow-up period and will be done by a single calibrated examiner
  The PI will be evaluated by using Silness-Loe PI (0 = no plaque, 1 = thin film of plaque along the gingival margin, 2 = Moderate accumulation of plaque in the sulcus, 3 = Large amount of plaque in sulcus along the gingival margin).
Probing pocket depth (PPD) change from baseline to 6 months | PPD will be taken at baseline, 1 month, 3 months and 6months after the intervention during the follow-up period and will be done by a single calibrated examiner.
  The PPD will be clinically measured by using UNC 15 periodontal probe from the gingival margin to the depth of the pocket. An individually customized positioning stent will be fabricated for each patient to ensure accuracy and reproducibility of the measurements.
Gingival recession (GR) change from baseline to 6 months | GR will be taken at baseline, 1 month, 3 months and 6months after the intervention during the follow-up period and will be done by a single calibrated examiner.
  The GR will be clinically measured by using UNC 15 periodontal probe from the CEJ to the gingival margin.
Bleeding on probing (BoP) change from baseline to 6 months | BoP will be taken at baseline, 1 month, 3 months and 6months after the intervention during the follow-up period and will be done by a single calibrated examiner.
  The BoP will be clinically measured by using UNC 15 periodontal probe from the CEJ to the gingival margin.
Postoperative Pain | Postoperative Pain will be measured after the surgical procedure and 2 weeks post-surgical.
  Postoperative Pain will be measured by using visual analogue score (0-10).
Patient satisfaction | Patient satisfaction will be measured 2 weeks post-surgical.
  Patient satisfaction will be measured using a survey.

CONTACTS AND LOCATIONS:
Overall Officials: Ghada M. Abouhussein, Bachelor, Principal Investigator — Cairo University; Weam El-Battawy, Ass professor, Study Director — Cairo University; Nesma Shemais, Ass lecturer, Study Chair — Cairo University
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Egypt